CLINICAL TRIAL: NCT05861882
Title: THE CORRELATİON BETWEEN FUNCTIONAL MOVEMENT ANALYSIS AND CORE STABILISATION AND Y BALANCE TEST IN HANDBALL PLAYERS
Brief Title: ASSESSMENT OF THE HANDBALL PLAYERS
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, THE CORRELATİON BETWEEN FUNCTIONAL MOVEMENT ANALYSIS AND CORE STABILISATION AND Y BALANCE TEST IN HANDBALL PLAYERS, Kırıkkale University
Other Study IDs: Gurbuz01
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Functional Movement Disorder; Sport Injury
Keywords: functional movement screen, balance, core stabilization, sport injury
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- handball player: * To be a licensed handball athlete
  * Not having undergone a surgical operation involving the musculoskeletal system in the last six months
  * Not having any obstacle to perform the tests to be performed within the study
  * Volunteering to participate in the study
  Interventions: Other: functional movement screen; Other: survey application; Other: Y balance test; Other: Core stabilization assessment
- sedantary young people: -being a volunteer
  Interventions: Other: functional movement screen; Other: survey application; Other: Y balance test; Other: Core stabilization assessment

INTERVENTIONS:
Other: functional movement screen — FMS consists of seven test component which are used to evaluate various main movement models.Individuals completed one by one deep squat, high stepping, single line lunge, shoulder mobility, straight leg raises, trunk stability push-ups, rotation stability which are component tests. Subcomponent tests assess asymmetry by measuring the individual bilaterally. Each component test was scored on an ordinal scale (0 to 3 points), with a maximum score of 3, based on the quality of the movement. Less than 3 points indicated that the individual performed some form of compensation or was unable to complete the entire movement.While individuals were doing these tests, they were recorded in the video , the final scoring was done by evaluating the images. The scores of the component tests were summed, resulting in a composite score between 0 and 21 points, with a maximum score of 21
Other: survey application — Participants are evaluated with kasari physical activity survey. According to the FIT score, physical activity level is commented as sedentary between 0-20, poor between 21-40, normal between 41-60, good between 61-80 and perfect between 81-100
Other: Y balance test — YBT, which is performed in the standing position on one leg , is dynamic a test. Participants stood on the footplate in the centre of the Y Balance Test area and then, it was given instruction them that they should maintain a single leg stance while reaching as far as possible with the opposite leg and return to the starting position on the centre platform without losing balance.In the test, individuals were asked to reach the maximum distance in 3 directions (anterior, posteromedial and posterolateral), allowing 3 trials for each leg. The maximum reach distance was recorded for each consecutive trial
Other: Core stabilization assessment — The flexor muscle endurance test is initiated with the subject in a sitting position, with the back leaning against an apparatus angled 60 degrees from the floor. Both knees and hips are flexed to 90 degrees and the support apparatus is withdrawn and the time the person maintains the position is recorded The extensor muscle endurance test is performed with the upper trunk extended towards the end of the bed on which the test is performed and the pelvis, knees and hips fixed. The time the upper trunk maintains its level is recorded The lateral bridge test was performed with the individual lying in the full side bridge position (left and right side separately). Individuals supported themselves on one elbow and their feet while lifting their hips off the floor to form a straight line from head to toe. The test was terminated when the individual lost the straight back posture and/or their hips touched the floor.

SUMMARY:
''This study aims to determine the relationship between functional movement screen (FMS), core stabilization and Y balance test. The study will include evaluations on 30 handball players and 30 sedentary individuals.'' Functional movement analysis is a biomechanical screening and evaluation system to identify limitations and asymmetries in 7 basic movements. This system reveals the kinetic chain interaction between mobility and stability required for basic performance. Unlike conventional assessment methods, FHA focuses on the efficiency and quality of the movement pattern, not on the number of repetitions or weight lifted.

The main aim of the study was to reveal the relationship between functional movement screen and core endurance and Y balance test evaluations in handball players with objective data. Functional movement is the general name of the activities performed by individuals for function and the movements performed by individuals for function are examined with analysis methods. In an effective analysis, if people do not have appropriate stability and mobility, it is determined from which muscle-muscle group or joint the problem originates. Analyses play a role in determining which of the stabilization, mobilization and flexibility factors are problematic at which stage of the function. In addition, these methods are effective in preventing possible injuries while helping to improve balance, strength and power characteristics of individuals. Core stabilization problems cause significant posture and stabilization problems. These problems are reflected in functional movements. Core stabilization problems are thought to have negative effects on functional movement analysis scores. Active athletes with this problem will be more affected. This study also aimed to observe the differences between athletes and sedentary individuals.

Studies defined the core as the part of the body in the musculoskeletal system consisting of the proximal lower extremities, abdominal structures, hips, pelvis and spine and stated that the core muscles are composed of the trunk and pelvis muscles. It is argued that trunk and pelvis stabilization is essential for all movements of the extremities. The transversus abdominis and multifidus work in cocontraction and control excessive anterior pelvic tilt, which is known to be associated with femoral internal rotation and adduction. The musculature of the core is referred to as the muscular corset over the trunk and spine that stabilizes the body with or without limb movement. The strength and stabilization of the core affects the fitness and physical fitness of athletes. Core exercises should be included in exercise programs planned to improve athletic performance. Core endurance tests have been defined to reveal the relationship between core stabilization and performance. Lateral bridge test and trunk flexor test are the preferred core endurance tests in this study. The Y balance test is a dynamic test that requires strength, flexibility, core control and proprioception in a single-legged stance. Functional movement analysis, core stabilization tests and Y balance test are assessment scales that provide objective data on stabilization, postural alignment and spinal alignment. It is envisaged that these three assessment parameters will support each other after the study.

Functional movements are widely used during both daily and sports activities. Core stabilization and dynamic balance are the factors that determine the quality of functional movements. These movements become more important for athletes as they affect their sporting success. Athletes need a good evaluation to ensure and maintain success. Since handball is defined as a sport that requires a lot of effort, the risks increase and it becomes clear that the evaluation should be done with a holistic approach.Injuries in handball develop due to multifactors.Biomechanical, kinesthetic and functional losses in players should be determined to prevent injuries.Functional movement analysis, core stabilization, Y balance test will give us detailed information about posture, limb alignment and asymmetry, spinal smoothness, dynamic balance and will give us the chance to analyze whether there is a correlation between these tests.

DETAILED DESCRIPTION:
In this study, it will be questioned whether functional movement analysis can be considered as a part of core stabilization assessment in sedentary and athletes. The effects of dynamic balance on functional activity will be observed. It is aimed to evaluate the relationship between the test results and injury risks in the individuals participating in the study and what the most accurate exercises can be according to the evaluation parameters of the person to prevent injuries.

This study includes the first evaluations of fms in a young age group. It will be a pilot study in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed handball athlete
* Not having undergone a surgical operation involving the musculoskeletal system in the last six months
* Not having any obstacle to perform the tests to be performed within the study
* Volunteering to participate in the study

Exclusion Criteria:

* Feeling any discomfort during the tests
* Not wanting to continue working

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 young people licensed by the Turkish Handball Federation handball players and 30 sedentary young volunteers participated.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
FUNCTİONAL MOVEMENT SCREEN | 1 day
  FMS consists of seven test component which are used to evaluate various main movement models.Individuals completed one by one deep squat, high stepping, single line lunge, shoulder mobility, straight leg raises, trunk stability push-ups, rotation stability which are component tests. Subcomponent tests assess asymmetry by measuring the individual bilaterally. Each component test was scored on an ordinal scale (0 to 3 points), with a maximum score of 3, based on the quality of the movement. Less than 3 points indicated that the individual performed some form of compensation or was unable to complete the entire movement.While individuals were doing these tests, they were recorded in the video , the final scoring was done by evaluating the images. The scores of the component tests were summed, resulting in a composite score between 0 and 21 points, with a maximum score of 21

SECONDARY OUTCOMES:
Y BALANCE TEST | 1 day
  YBT, which is performed in the standing position on one leg , is dynamic a test. Participants stood on the footplate in the centre of the Y Balance Test area and then, it was given instruction them that they should maintain a single leg stance while reaching as far as possible with the opposite leg and return to the starting position on the centre platform without losing balance.In the test, individuals were asked to reach the maximum distance in 3 directions (anterior, posteromedial and posterolateral), allowing 3 trials for each leg. The maximum reach distance was recorded for each consecutive trial
CORE STABİLİZATİON ASSESMENT | 1 day
  The flexor muscle endurance test is initiated with the subject in a sitting position, with the back leaning against an apparatus angled 60 degrees from the floor. Both knees and hips are flexed to 90 degrees and the support apparatus is withdrawn and the time the person maintains the position is recorded.
  The extensor muscle endurance test is performed with the upper trunk extended towards the end of the bed on which the test is performed and the pelvis, knees and hips fixed. The time the upper trunk maintains its level is recorded.
  The lateral bridge test was performed with the individual lying in the full side bridge position (left and right side separately). Individuals supported themselves on one elbow and their feet while lifting their hips off the floor to form a straight line from head to toe. The test was terminated when the individual lost the straight back posture and/or their hips touched the floor.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No